CLINICAL TRIAL: NCT06426563
Title: Microwave Ablation Versus Radiofrequency Ablation for the Treatment of Moderate-sized Benign Thyroid Nodules, a Randomized Controlled Trial
Brief Title: MWA vs RFA for the Treatment of Moderate-sized Benign Thyroid Nodules
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Man Him Matrix Fung, Clinical Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UW 24-141
Record Dates: First submitted 2024-05-17; First posted 2024-05-23 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Thyroid Nodule (Benign); Ablation Therapy
Keywords: Ablation therapy; Thyroid nodule; benign; RFA; MWA
MeSH Terms: conditions — Thyroid Nodule

STUDY DESIGN:
Intervention Model Description: One group is for radiofrequency ablation treatment (RFA), another group is for microwave ablation treatment (MWA)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiofrequency ablation treatment (RFA) to thyroid nodule (Active Comparator): Participants who are undergo thyroid nodule treatment by RFA
  Interventions: Procedure: Ablation treatment of thyroid nodule
- Microwave ablation treatment (MWA) to thyroid nodule (Active Comparator): Participants who are undergo thyroid nodule treatment by MWA
  Interventions: Procedure: Ablation treatment of thyroid nodule

INTERVENTIONS:
Procedure: Ablation treatment of thyroid nodule — Use Radiofrequency or Microwave ablation device to treat thyroid nodule

SUMMARY:
Thyroid nodule is a common condition that affects up to 60% of the population. There is an estimated 10% lifetime probability of developing a thyroid nodule. Although most thyroid nodules are benign, up to 10-15% can enlarge to cause compressive symptoms including neck pressure and discomfort, dysphagia, dyspnea, and dysphonia. The conventional treatment for these benign but problematic nodules has been thyroidectomy. Although generally a low risk operation, thyroidectomy is associated with some risk for recurrent laryngeal nerve injury, bleeding, infection, and need for thyroid hormone supplementation. Since the early 2000s, ultrasound-guided percutaneous thermal ablation has emerged as a potential alternative treatment to surgery for benign thyroid nodules. Of the myriad ablation methods, the most commonly used techniques are radiofrequency ablation (RFA) and microwave ablation (MWA). [1-3] A growing body of evidence shows that RFA is an effective treatment for benign solid thyroid nodules, toxic adenomas, and thyroid cysts resulting in overall volume reduction ranges of 40-80% at 1 year, with durable resolution of compressive and hyperthyroid symptoms. However, RFA is not without its limitations. Radiofrequency waves can be limited by the heat sink effect and tissue char leading to longer procedure times and potentially less optimal outcomes in larger, hypervascular, and/or more cystic nodules.

Microwave ablation (MWA) is another ablative technique that uses electromagnetic energy waves to cause tissue hyperthermia and coagulative necrosis. It generally causes higher ablation temperatures than RFA and is less subject to the heat sink effect, and therefore can facilitate more efficient ablation procedures. Current evidence comparing RFA versus MWA for thyroid ablation was limited and was either retrospective, non-randomized [4-9], under-powered, or with an unequal baseline. The results from these studies were also conflicting, suggesting suboptimal quality of evidence and bias due to non-standardized technique of ablation across studies. To date, there is no randomized controlled trial comparing the efficacy and safety of RFA versus MWA for the treatment of benign thyroid nodules. Given the higher ablation temperatures, freedom from heat sink effect, and no influence from impedance changes during ablation, MWA may achieve different treatment efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients >/=18 years of age
2. Nodule maximal diameter ≥2cm and nodule volume <20ml
3. Nodule being predominantly solid (≥80% solid)
4. Confirmed benign nature of nodules, either by : two benign fine needle biopsies, with the most recent biopsy performed within 1 year of enrollment in study or one benign fine needle biopsy and low suspicion characteristics on ultrasound
5. Both functional and non-functional nodules are eligible.

Exclusion Criteria:

1. Cytologically indeterminate nodules
2. Nodules with substernal extension or posterior extension that cannot be viewed sufficiently with ultrasound
3. current pregnancy or cardiac arrhythmias; presence of pacemaker or any medical condition that renders patient unfit for thermal ablation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
To measure the volume reduction ratio (VRR) of the first ablated nodule at each procedure at 12-months post-procedure | 12 months

SECONDARY OUTCOMES:
To measures nodule recurrence rate | 12-24 months
To measures thyroid nodule regrowth rate | 12-24 months
To measure cosmetic score by investigator (1-4) | 12-24 months
  To measure cosmetic score from 1 to 4 (1 is No palpable goitre, 2 is Palpable goitre but invisible, 3 is Goitre only visible to experienced clinician, 4 is Easily visible goitre)
To measure the compressive symptom scores (from 0 - 100) | 12-24 months
  compressive symptom score from 0 (no compression feeling) to 100 (the most compressive)
To measure swallowing impairment scores by questionnaire (SIS-6) | 12-24 months
  Swallowing Impairment Index (SIS-6) is an assessment tool about swallowing dysfunction and symptom. It comprises six question items ranging from 0 (no impairment) to 24 (maximum impairment)
To measure pain score (0-10) after ablation treatment | 12-24 months
  0 is no pain, 10 is the most painful
Change of quality of life by SF12 ver 2 | 12-24 months
  SF-12(v2) is an assessment tool about quality of life. It comprises 12 question items ranging from 11 (worst quality of life) to 56 (best quality of life).

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lang BHH, Fung MMH. Safety and Efficacy of Single-Session Radiofrequency Ablation Treatment for Benign Non-toxic Multinodular Goiter. World J Surg. 2022 Jul;46(7):1704-1710. doi: 10.1007/s00268-022-06527-8. Epub 2022 Mar 21. PMID 35313358
- [Background] Cheng Z, Che Y, Yu S, Wang S, Teng D, Xu H, Li J, Sun D, Han Z, Liang P. US-Guided Percutaneous Radiofrequency versus Microwave Ablation for Benign Thyroid Nodules: A Prospective Multicenter Study. Sci Rep. 2017 Aug 25;7(1):9554. doi: 10.1038/s41598-017-09930-7. PMID 28842651
- [Background] Wu W, Gong X, Zhou Q, Chen X, Chen X. Ultrasound-Guided Percutaneous Microwave Ablation for Solid Benign Thyroid Nodules: Comparison of MWA versus Control Group. Int J Endocrinol. 2017;2017:9724090. doi: 10.1155/2017/9724090. Epub 2017 Nov 23. PMID 29333159
- [Background] He L, Zhao W, Xia Z, Su A, Li Z, Zhu J. Comparative efficacy of different ultrasound-guided ablation for the treatment of benign thyroid nodules: Systematic review and network meta-analysis of randomized controlled trials. PLoS One. 2021 Jan 20;16(1):e0243864. doi: 10.1371/journal.pone.0243864. eCollection 2021. PMID 33471820
- [Background] Hu K, Wu J, Dong Y, Yan Z, Lu Z, Liu L. Comparison between ultrasound-guided percutaneous radiofrequency and microwave ablation in benign thyroid nodules. J Cancer Res Ther. 2019;15(7):1535-1540. doi: 10.4103/jcrt.JCRT_322_19. PMID 31939434
- [Background] Guo DM, Chen Z, Zhai YX, Su HH. Comparison of radiofrequency ablation and microwave ablation for benign thyroid nodules: A systematic review and meta-analysis. Clin Endocrinol (Oxf). 2021 Jul;95(1):187-196. doi: 10.1111/cen.14438. Epub 2021 Mar 2. PMID 33556187
- [Background] Jin H, Fan J, Lu L, Cui M. A Propensity Score Matching Study Between Microwave Ablation and Radiofrequency Ablation in Terms of Safety and Efficacy for Benign Thyroid Nodules Treatment. Front Endocrinol (Lausanne). 2021 Mar 9;12:584972. doi: 10.3389/fendo.2021.584972. eCollection 2021. PMID 33767666
- [Background] Kim JH, Baek JH, Lim HK, Ahn HS, Baek SM, Choi YJ, Choi YJ, Chung SR, Ha EJ, Hahn SY, Jung SL, Kim DS, Kim SJ, Kim YK, Lee CY, Lee JH, Lee KH, Lee YH, Park JS, Park H, Shin JH, Suh CH, Sung JY, Sim JS, Youn I, Choi M, Na DG; Guideline Committee for the Korean Society of Thyroid Radiology (KSThR) and Korean Society of Radiology. 2017 Thyroid Radiofrequency Ablation Guideline: Korean Society of Thyroid Radiology. Korean J Radiol. 2018 Jul-Aug;19(4):632-655. doi: 10.3348/kjr.2018.19.4.632. Epub 2018 Jun 14. PMID 29962870
- [Background] Huh JY, Baek JH, Choi H, Kim JK, Lee JH. Symptomatic benign thyroid nodules: efficacy of additional radiofrequency ablation treatment session--prospective randomized study. Radiology. 2012 Jun;263(3):909-16. doi: 10.1148/radiol.12111300. Epub 2012 Mar 21. PMID 22438360
- [Background] Lim HK, Lee JH, Ha EJ, Sung JY, Kim JK, Baek JH. Radiofrequency ablation of benign non-functioning thyroid nodules: 4-year follow-up results for 111 patients. Eur Radiol. 2013 Apr;23(4):1044-9. doi: 10.1007/s00330-012-2671-3. Epub 2012 Oct 25. PMID 23096937